CLINICAL TRIAL: NCT00794729
Title: Sub-Study Evaluating the Quality of Different Methods of Obtaining Informed Consent"
Brief Title: Evaluating the Quality of Different Methods of Obtaining Informed Consent
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909011; 09-CC-N011
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-14

CONDITIONS: Healthy Volunteers; Participant Satisfaction
Keywords: Healthy Volunteers; Consents

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a sub-study of a drug development study conducted by Pfizer, Inc. It will evaluate how well people who participate in research studies understand from the study consent form what the purpose of the study is, the risks and benefits of participating, the procedures they will undergo and their right to withdraw from the study before it ends. It will compare the understanding and satisfaction of those who are given a standard consent form with those who are given a simpler, concise consent form and examine how their understanding of the information is affected by the length, complexity, format, and reading level of the document.

People 18 years of age and older who are participating in a Pfizer drug development study and who are able to read and write English may be eligible for this sub-study.

Participants in Pfizer's drug development study who agree to participate in this sub-study are randomized to receive either the standard consent form or the concise consent form. The standard consent consists of a detailed, multiple page consent form. The concise form is simpler, written at a lower reading comprehension level. Both forms contain all of the required elements of informed consent according to federal regulations, and include information needed to make a decision about participating in the study. Each form also contains information regarding participation in this sub-study. The standard group signs the standard consent form; the concise group is given the standard consent after reviewing the concise form and is asked to review and sign it.

After reviewing the consent form for the main study, participants complete a 20-minute questionnaire that includes questions that measure understanding of study information such as its purpose, risks and benefits, compensation schemes, and other information. Additional questions ask about how the participants made the decision to enroll in the study.

...

DETAILED DESCRIPTION:
This informed consent study is a sub-study of phase 1 drug development studies conducted by Pfizer International and is designed to evaluate research participant understanding and satisfaction after being randomized to receive written study information from either a standard consent form or a concise consent form.

ELIGIBILITY:
* INCLUSION CRITERIA:

All willing adults at least 18 years old who come to the Pfizer CRU to consider volunteering for a phase 1 study for which there is a consent sub-study and who are able to read and answer questions in English are eligible to participate in the sub-study. Only adults (over 18 years old) who can provide their own consent will be included. Because the consent forms for Pfizer studies are written in English, the sub-study will only include individuals who can read and answer questions in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-10-16; Study Completion 2011-09-14

CONTACTS AND LOCATIONS:
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Background] Sugarman J, McCrory DC, Powell D, Krasny A, Adams B, Ball E, Cassell C. Empirical research on informed consent. An annotated bibliography. Hastings Cent Rep. 1999 Jan-Feb;29(1):S1-42. No abstract available. PMID 10051999
- [Background] Edwards SJ, Lilford RJ, Thornton J, Hewison J. Informed consent for clinical trials: in search of the "best" method. Soc Sci Med. 1998 Dec;47(11):1825-40. doi: 10.1016/s0277-9536(98)00235-4. PMID 9877351
- [Background] Bergler JH, Pennington AC, Metcalfe M, Freis ED. Informed consent: how much does the patient understand? Clin Pharmacol Ther. 1980 Apr;27(4):435-40. doi: 10.1038/clpt.1980.60. PMID 6987027